CLINICAL TRIAL: NCT06288945
Title: Effect of an Educational Program on Health-related Outcomes of Patients With Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Emad Rabie, Lecturer, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dry eye syndrome
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The educational nursing interventions were individually administered to each participant in the study group in two sessions which were conducted after the assessment phase on the day of the eye examination at the ophthalmology outpatient clinic and after the diagnosis of dry eye syndrome.
  Interventions: Other: Educational Program
- Control Group (No Intervention): The control group was selected first and did not receive the educational program for dry eye syndrome

INTERVENTIONS:
Other: Educational Program — The educational program included information about definition and causes of Dry eye syndrome (DES), symptoms of DES, diagnostic measures of DES, differentiation between DES and eye allergy, complications of DES, the effect of DES on vision, management of DES, health education about proper eyelid hygiene, proper nutrition to improve the quality of tear film, measures, and precautions to prevent DES such as avoiding exposure to smoke and environmental changes, avoiding prolonged periods in air-conditioned environments; limiting contact lens use to shorter periods, avoiding staring at the computer screen or smartphone for long periods, and taking frequent breaks. In addition, health education about the importance of compliance with the treatment of DES, and instructions to maintain normal eye and vision in patients with DES.
  Arms: Study Group

SUMMARY:
Dry eye syndrome (DES) is a widespread ocular disease affecting the general population. It is a complex disorder affecting the surface of the eye, marked by an imbalance in the tear film and ocular symptoms. Therefore this study was done to determine the effect of an educational program on health-related outcomes of patients with DES including the severity of symptoms related to DES and their influence on visual-related functions

DETAILED DESCRIPTION:
Dry eye syndrome (DES) is a prevalent chronic, inflammation resulting in eye discomfort, irritation, tiredness, and visual abnormalities that can make it difficult to read, use a computer, drive, or engage in other activities (1). It represents a set of tears film disorders caused by decreased tears formation or increased tears evaporation; it causes visual symptoms, ocular surface inflammation, and discomfort. In addition, DES leads to impaired visual function and can negatively affect the outcomes of cataract surgery (2).Therefore this study was done to determine the effect of an educational program on health-related outcomes of patients with DES including the severity of symptoms related to DES and their influence on visual-related functions

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 60 years old.
* Alert, and able to communicate.

Exclusion Criteria:

* patients with recent ocular surgeries in the last 3 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
ocular irritation symptoms associated with Dry eye syndrome and their effect on functions related to vision | 8 months
  Ocular surface disease index (OSDI) was developed by the Outcomes Research Group at Allergan Inc in 1997 (20). It is a 12-item questionnaire developed to assess ocular irritation symptoms associated with dry eye syndrome and their effect on functions related to vision.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria university, Alexandria, Egypt

REFERENCES:
- [Background] Al-Mohtaseb Z, Schachter S, Shen Lee B, Garlich J, Trattler W. The Relationship Between Dry Eye Disease and Digital Screen Use. Clin Ophthalmol. 2021 Sep 10;15:3811-3820. doi: 10.2147/OPTH.S321591. eCollection 2021. PMID 34531649
- [Background] Akpek EK, Amescua G, Farid M, Garcia-Ferrer FJ, Lin A, Rhee MK, Varu DM, Musch DC, Dunn SP, Mah FS; American Academy of Ophthalmology Preferred Practice Pattern Cornea and External Disease Panel. Dry Eye Syndrome Preferred Practice Pattern(R). Ophthalmology. 2019 Jan;126(1):P286-P334. doi: 10.1016/j.ophtha.2018.10.023. Epub 2018 Oct 23. No abstract available. PMID 30366798
- [Derived] Rabie EAEGA, ElRazkey JY, Ahmed HA. Empowering vision: the impact of nursing-led educational program on patients with dry eye syndrome. BMC Nurs. 2024 Sep 27;23(1):693. doi: 10.1186/s12912-024-02318-9. PMID 39334075